CLINICAL TRIAL: NCT02233738
Title: Group Motivational Interviewing (GMI) For Homeless Veterans In VA Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 13-317
Record Dates: First submitted 2014-08-21; First posted 2014-09-08 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Alcoholism; Substance-related Disorders; Dual Diagnosis
Keywords: Alcoholism; Substance-related disorders; Dual Diagnosis
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Motivational Interviewing (GMI) (Experimental): Group Motivational Interviewing (GMI) participants will receive four structured, back-to-back, 90-min sessions consistent with the central principles and spirit of Motivational Interviewing (MI). GMI, which is based on a manualized protocol, is specifically designed for dually diagnosed Veterans. A focus of the intervention creates awareness of the relationship between the substance use and co-existing psychiatric disorder and the importance of treating both.
  Interventions: Behavioral: Group Motivational Interviewing (GMI)
- Control Treatment Condition (CT) (Active Comparator): Control Treatment Condition (CT): Participants in CT will attend four sessions equal in time and length to Group Motivational Interviewing (GMI) (i.e., 90 minutes) and will involve the following topics: A popular 'box activity': participants will anonymously write evocative questions on slips of paper involving their personal concerns that are placed in a box and, when randomly selected, opened for group discussion (e.g., "How do I talk to my family about my alcohol problem?"), money management with feedback (2 sessions), and cooking-home maintenance.
  Interventions: Behavioral: Control Treatment Condition (CT)

INTERVENTIONS:
Behavioral: Group Motivational Interviewing (GMI) — Participants randomized to Group Motivational Interviewing (GMI) will receive four structured, back-to-back, 90-minute sessions consistent with the central principles and spirit of Motivational Interviewing (MI). GMI, which is based on a manualized protocol, is specifically designed for dually diagnosed Veterans. A focus of the intervention creates awareness of the relationship between the substance use and co-existing psychiatric disorder and the importance of treating both.
  Arms: Group Motivational Interviewing (GMI)
Behavioral: Control Treatment Condition (CT) — Control Treatment Condition (CT): Participants in CT will attend four sessions equal in time and length to GMI (i.e., 90 minutes) and will involve the following topics: A popular 'box activity': participants will anonymously write evocative questions on slips of paper involving their personal concerns that are placed in a box and, when randomly selected, opened for group discussion (e.g., "How do I talk to my family about my alcohol problem?"), money management with feedback (2 sessions), and cooking-home maintenance.
  Arms: Control Treatment Condition (CT)

SUMMARY:
Homeless Veterans with substance use disorders (SUDs) are a major group served by VA and are heavily represented in VA housing. VA recently adopted a 'Housing First' approach emphasizing rapid housing placement to initiate recovery without requiring sobriety and will necessitate SUD interventions that are efficient and easily layered onto existing services. The proposed study will investigate the effectiveness, implementation process, and cost estimate of Group Motivational Interviewing (GMI) for Veterans with SUDs in VA housing (Housing Urban Development-VA Support Housing [HUD-VASH] and Grant and per Diem [GPD]). Outcomes will be assessed at multiple time points using a multi-modal approach. The ultimate goal of this research is to establish the basis of a GMI dissemination and implementation course of action for highly vulnerable homeless Veterans in VA housing for achieving their greatest success in attaining housing stability.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans Health Care:

VA set an ambitious goal for ending homelessness among Veterans by 2015. Housing Urban Development-VA Support Housing [HUD-VASH] and Grant and per Diem [GPD] are two primary VA housing programs to help Veterans exit homelessness. Substance abuse among Veterans in VA housing is a major risk factor for worsening psychopathology and housing instability. Despite recent adoption of a Housing First approach, many VA housing programs lack the staff infrastructure to manage substance use disorders (SUDs). This is a significant problem as 60% (conservative estimate) of Veterans in VA housing have SUDs and these Veterans show greater psychopathology compared to their counterparts without SUDs. These issues warrant substantial need for SUD programs in VA housing that are efficient to deploy, easily layered onto existing services, and require minimal staff to operate. The current study addresses this current void in VA treatment services in that it investigates the effectiveness, implementation process, and cost estimate of treatment of an adaptation of motivational interviewing, an empirically supported intervention with strong impact on reducing substance use and enhancing treatment engagement, in a group format, referred to as Group Motivational Interviewing (GMI) for Veterans with SUDs in VA housing. Data from this project, if shown to be promising, will establish the basis of a GMI dissemination and implementation course of action for highly vulnerable homeless Veterans in VA housing for achieving their greatest success in attaining housing stability.

Background:

There is a significant need for 'wraparound' treatment services in VA housing for addressing SUDs. Homeless Veterans with SUDs are vulnerable to treatment dropout, rendering them susceptible to relapse, while their continuation in outpatient care during their participation in VA housing leads to improved clinical outcomes. According to systematic reviews, individual motivational interviewing reduces the incidence of substance use disorders, when compared to no treatment, but is labor intensive. As VA moves toward a 'Housing First' paradigm where greater numbers of homeless Veterans will continue to use substances while in VA housing, delivery of GMI (which may be less labor intensive) to these patients will be important for initiating and maintaining their recovery as well as enhancing their psychosocial integration and quality of life. In a prior controlled trial conducted by the Principal Investigator, GMI resulted in significantly higher outpatient treatment engagement and lower substance use compared to treatment-as-usual among dually diagnosed Veterans.

Objectives:

Study objectives are consistent with VA housing recommendations focusing on patient recovery, health services promotion, and treatment implementation evaluation. GMI will be compared to a control treatment condition (CT) on (Specific Aim I; Five outcomes: (Primary Hypothesis 1): treatment engagement; (Primary Hypothesis 1): substance use; (Secondary H2): psychosocial integration (e.g., social support, community participation); (Secondary H3) quality of life/psychiatric indices; and (Secondary H4): number of days engaging in structured/productive work activities in the 6-month follow up. Specific Aim II involves a process evaluation for documenting (A) formative (e.g., developmental), (B) process, and (C) summative outcomes; and Specific Aim III involves estimation of cost of intervention in terms of direct costs, indirect costs of staff, costs of capital and workload measures for future implementation and dissemination research.

Methods:

Randomized controlled trial comparing GMI to control treatment (CT) across five critical outcomes. 186 Veterans in VA housing services (93 per treatment arm) will be enrolled with a diagnosis of alcohol or drug abuse/dependence. Recruitment will take place in Charleston VA Medical Center HUD-VASH & GPD. Participants will be randomly assigned to (1) GMI or (2) CT, each consisting of 4 sessions, and will be evaluated at 1, 3, and 6 months. Participants with a non-substance related DSM-V disorder (e.g., major depressive disorder, PTSD) will be eligible for the study. Analyses will be conducted using generalized linear mixed models (GLMM) approach.

Significance to Veterans:

Homeless Veterans with SUDs represent one of the largest and most chronic groups of psychiatric patients treated in the VA Healthcare System. With the ongoing execution of VA's "Plan to End Veteran Homelessness," Veterans entering housing require interventions that can be feasibly implemented with minimal reorganization of existing services. GMI is based on motivational interviewing, an empirically valid treatment that aligns with Veteran-centered recovery models including Harm Reduction and more traditional treatment philosophies. The investment in GMI for VA housing may be minimal as it requires only a few staff to operate in relatively short time (e.g., 4 sessions, 90-min each) with modest (20 hours) staff training. It can be layered onto existing services with little interruption or reorganization of staff, and it has potential to be offered to larger numbers of Veterans with SUDs in VA housing who would otherwise not receive this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women Veterans currently in Housing Urban Development-VA Support Housing [HUD-VASH] and Grant and per Diem [GPD]), newly entering the program but not yet housed, or Veterans on the HUD-VASH interest (wait) list.
* Able to comprehend English.
* Meets DSM-V criteria for a current substance use disorder and have used substances in the 30 days prior to treatment entry. Participants on medications targeting their substance use must be stabilized on medications for at least 2 weeks before therapy initiation.
* May meet criteria a mood, anxiety or other psychiatric disorder. Participants on maintenance medications for a mood or anxiety disorder must be stabilized on medications for at least 2 weeks before therapy initiation.
* Able to adequately provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Willing to commit to 4 group therapy sessions, baseline, 1, 3, and 6 month follow-up assessments.

Exclusion Criteria:

* Active suicidal or homicidal ideation with a plan as this is likely to require hospitalization or other interventions that could interfere with study participation.
* Unstable psychiatric condition that is likely to require hospitalization or other interventions that would interfere with study participation.
* Unstable medical condition or one that may require hospitalization during the course of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Santa Ana, PhD MA BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jaconis M, Santa Ana EJ, Killeen TK, Badour CL, Back SE. Concurrent treatment of PTSD and alcohol use disorder via telehealth in a female Iraq veteran. Am J Addict. 2017 Mar;26(2):112-114. doi: 10.1111/ajad.12481. Epub 2017 Jan 24. PMID 28118514
- [Result] Gebregziabher M, Voronca D, Teklehaimanot A, Santa Ana EJ. Weibull mixture regression for marginal inference in zero-heavy continuous outcomes. Stat Methods Med Res. 2017 Jun;26(3):1476-1499. doi: 10.1177/0962280215583402. Epub 2015 Apr 22. PMID 25902801
- [Result] Shorey RC, Martino S, Lamb KE, LaRowe SD, Santa Ana EJ. Change talk and relatedness in group motivational interviewing: a pilot study. J Subst Abuse Treat. 2015 Apr;51:75-81. doi: 10.1016/j.jsat.2014.11.003. Epub 2014 Nov 20. PMID 25488505
- [Result] Santa Ana EJ, LaRowe SD, Armeson K, Lamb KE, Hartwell K. Impact of group motivational interviewing on enhancing treatment engagement for homeless Veterans with nicotine dependence and other substance use disorders: A pilot investigation. Am J Addict. 2016 Oct;25(7):533-41. doi: 10.1111/ajad.12426. Epub 2016 Sep 2. PMID 27589072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 481 patients screened between September 2015 and January 2018, 38% (n=185) were consented and enrolled. However, only 184 participants were randomized because 1 withdrew during baseline assessments.
Groups:
- Control Treatment Condition (CT): Control Treatment Condition (CT): Participants in CT will attend four sessions equal in time and length to GMI (i.e., 90 minutes) and will involve the following topics: A popular 'box activity', participants will anonymously submit questions on involving their personal concerns that are placed in a box and, when randomly selected, opened for group discussion money management with feedback (2 sessions), cooking-home maintenance, and psycho-education about substance use.
Period: Overall Study
Arm/Group | Group Motivational Interviewing (GMI) | Control Treatment Condition (CT)
Started | 93 | 91
1 Month Follow-Up | 89 | 82
3 Month Follow-Up | 87 | 77
6 Month Follow-Up | 85 | 75
Completed | 85 | 75
Not Completed | 8 | 16
Not completed — Lost to Follow-up | 5 | 12
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not return after Baseline | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Motivational Interviewing (GMI) | Control Treatment Condition (CT) | Total
Number analyzed (Participants) | 93 | 91 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.6) | 51.4 (9.5) | 51.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 87 | 87 | 174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 49 | 69 | 118
  Caucasian | 42 | 22 | 64
  Hispanic or Latino | 1 | 0 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 91 | 184

OUTCOME MEASURES:

1. Primary Outcome: Standard Ethanol Content Units (SECs) Baseline
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to baseline. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Unit
Groups:
- GMI - Standard Ethanol Content Units (SECs) at Baseline: GMI - Standard Ethanol Content Units (SECs) at Baseline
- LSEG - Standard Ethanol Content Units (SECs) at Baseline: LSEG - Standard Ethanol Content Units (SECs) at Baseline
Arm/Group | GMI - Standard Ethanol Content Units (SECs) at Baseline | LSEG - Standard Ethanol Content Units (SECs) at Baseline
Number analyzed (Participants) | 93 | 91
Standard Ethanol Content Unit | 179.9 [57.4 to 240.6] | 190.1 [68.5 to 244.7]

2. Primary Outcome: Standard Ethanol Content Units (SECs) at 1 Month
Description: The 1-month follow-up was conducted 30 days after day 1 of the treatment group. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to 1-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Standard Ethanol Content Units (SECs) at 1 Month: GMI - Standard Ethanol Content Units (SECs) at 1 month
- LSEG - Standard Ethanol Content Units (SECs) at 1 Month: LSEG - Standard Ethanol Content Units (SECs) at 1 month
Arm/Group | GMI - Standard Ethanol Content Units (SECs) at 1 Month | LSEG - Standard Ethanol Content Units (SECs) at 1 Month
Number analyzed (Participants) | 89 | 82
Standard Ethanol Content Units | 44.9 [0.0 to 28.2] | 36.9 [0.0 to 51.2]

3. Primary Outcome: Standard Ethanol Content Units (SECs) at 3 Months
Description: The 3-month follow-up was conducted 60 days after the 1-month follow-up. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days prior to 3-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Standard Ethanol Content Units (SECs) at 3 Months: GMI - Standard Ethanol Content Units (SECs) at 3 months
- LSEG - Standard Ethanol Content Units (SECs) at 3 Months: LSEG - Standard Ethanol Content Units (SECs) at 3 months
Arm/Group | GMI - Standard Ethanol Content Units (SECs) at 3 Months | LSEG - Standard Ethanol Content Units (SECs) at 3 Months
Number analyzed (Participants) | 87 | 77
Standard Ethanol Content Units | 50.1 [0.0 to 54.4] | 37.7 [0.0 to 44.5]

4. Primary Outcome: Standard Ethanol Content Units (SECs) at 6 Months
Description: The 6-month follow-up was conducted 90 days after the 3-month follow-up. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 90 days prior to 6-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents ALL standard drinks consumed within the stated time period.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Standard Ethanol Content Units (SECs) at 6 Months: GMI -Standard Ethanol Content Units (SECs) at 6 months
- LSEG - Standard Ethanol Content Units (SECs) at 6 Months: LSEG - Standard Ethanol Content Units (SECs) at 6 months
Arm/Group | GMI - Standard Ethanol Content Units (SECs) at 6 Months | LSEG - Standard Ethanol Content Units (SECs) at 6 Months
Number analyzed (Participants) | 85 | 75
Standard Ethanol Content Units | 96.5 [0.0 to 89.7] | 66.9 [0.0 to 104.4]

5. Primary Outcome: Peak SEC at Baseline
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to baseline. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed in a single day within the stated time period.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Peak SEC at Baseline: GMI - Peak SEC at Baseline
- LSEG - Peak SEC at Baseline: LSEG - Peak SEC at Baseline
Arm/Group | GMI - Peak SEC at Baseline | LSEG - Peak SEC at Baseline
Number analyzed (Participants) | 93 | 91
Standard Ethanol Content Units | 21.0 [12.0 to 25.6] | 19.1 [10.6 to 25.6]

6. Primary Outcome: Peak SEC at 1 Month
Description: The 1-month follow-up was conducted 30 days after day 1 of the treatment group. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to 1-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed on a single day within the stated time period.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Peak SEC at 1 Month: GMI - Peak SEC at 1 month
- LSEG - Peak SEC at 1 Month: LSEG - Peak SEC at 1 month
Arm/Group | GMI - Peak SEC at 1 Month | LSEG - Peak SEC at 1 Month
Number analyzed (Participants) | 89 | 82
Standard Ethanol Content Units | 4.8 [0.0 to 6.4] | 4.5 [0.0 to 7.4]

7. Primary Outcome: Peak SEC at 3 Months
Description: The 3-month follow-up was conducted 60 days after the 1-month follow-up. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days prior to 3-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed on a single day within the stated time period.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Peak SEC at 3 Months: GMI - Peak SEC at 3 months
- LSEG - Peak SEC at 3 Months: LSEG - Peak SEC at 3 months
Arm/Group | GMI - Peak SEC at 3 Months | LSEG - Peak SEC at 3 Months
Number analyzed (Participants) | 87 | 77
Standard Ethanol Content Units | 9.8 [0.0 to 13.0] | 5.9 [0.0 to 8.4]

8. Primary Outcome: Peak SEC at 6 Months
Description: The 6-month follow-up was conducted 90 days after the 3-month follow-up. The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 90 days prior to 6-month follow-up. Amount of alcohol consumption was converted to standard ethanol content units (SECs; or standard drinks) equivalent to 0.5 oz. of ethanol. This measure represents the most standard drinks consumed on a single day within the stated time period.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Standard Ethanol Content Units
Groups:
- GMI - Peak SEC at 6 Months: GMI - Peak SEC at 6 months
- LSEG - Peak SEC at 6 Months: LSEG - Peak SEC at 6 months
Arm/Group | GMI - Peak SEC at 6 Months | LSEG - Peak SEC at 6 Months
Number analyzed (Participants) | 85 | 75
Standard Ethanol Content Units | 10.3 [0.0 to 15.8] | 7.2 [0.0 to 10.8]

9. Primary Outcome: Alcohol Drink Days at Baseline
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to Baseline. This measure represents the number of days any alcohol was consumed within the stated time period.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: days
Groups:
- GMI -Alcohol Drink Days at Baseline: GMI - Alcohol Drink Days at Baseline
- LSEG - Alcohol Drink Days at Baseline: LSEG - Alcohol Drink Days at Baseline
Arm/Group | GMI -Alcohol Drink Days at Baseline | LSEG - Alcohol Drink Days at Baseline
Number analyzed (Participants) | 93 | 91
days | 13.3 [6.0 to 21.0] | 14.8 [8.0 to 21.0]

10. Primary Outcome: Alcohol Drink Days at 1 Month
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days after day 1 of the treatment group. This measure represents the number of days any alcohol was consumed within the stated time period.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Alcohol Drink Days at 1 Month: GMI - Alcohol Drink Days at 1 month
- LSEG - Alcohol Drink Days at 1 Month: LSEG - Alcohol Drink Days at 1 month
Arm/Group | GMI - Alcohol Drink Days at 1 Month | LSEG - Alcohol Drink Days at 1 Month
Number analyzed (Participants) | 89 | 82
Days | 4.6 [0.0 to 4.0] | 5.5 [0.0 to 5.0]

11. Primary Outcome: Alcohol Drink Days at 3 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days prior to 3-month follow-up. This measure represents the number of days any alcohol was consumed within the stated time period.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Alcohol Drink Days at 3 Months: GMI - Alcohol Drink Days at 3 months
- LSEG - Alcohol Drink Days at 3 Months: LSEG - Alcohol Drink Days at 3 months
Arm/Group | GMI - Alcohol Drink Days at 3 Months | LSEG - Alcohol Drink Days at 3 Months
Number analyzed (Participants) | 87 | 77
Days | 6.2 [0.0 to 9.5] | 6.6 [0.0 to 12.0]

12. Primary Outcome: Alcohol Drink Days at 6 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 90 days prior to 6-month follow-up. This measure represents the number of days any alcohol was consumed within the stated time period.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Alcohol Drink Days at 6 Months: GMI - Alcohol Drink Days at 6 months
- LSEG - Alcohol Drink Days at 6 Months: LSEG - Alcohol Drink Days at 6 months
Arm/Group | GMI - Alcohol Drink Days at 6 Months | LSEG - Alcohol Drink Days at 6 Months
Number analyzed (Participants) | 85 | 75
Days | 8.3 [0.0 to 13.7] | 8.3 [0.0 to 16.0]

13. Primary Outcome: Binge Drink Days at Baseline
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to Baseline. This measure represents the number of days the participant binge drank (5 or more standard drinks on a single day for males; 4 or more standard drinks on a single day for females).
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Binge Drink Days at Baseline: GMI - Binge Drink Days at Baseline
- LSEG - Binge Drink Days at Baseline: LSEG - Binge Drink Days at Baseline
Arm/Group | GMI - Binge Drink Days at Baseline | LSEG - Binge Drink Days at Baseline
Number analyzed (Participants) | 93 | 91
Days | 11.0 [4.0 to 19.0] | 12.0 [5.0 to 17.0]

14. Primary Outcome: Binge Drink Days at 1 Month
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to 1-month follow-up. This measure represents the number of days the participant binge drank (5 or more standard drinks on a single day for males; 4 or more standard drinks on a single day for females) within the stated time period.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Binge Drink Days at 1 Month: GMI - Binge Drink Days at 1 month
- LSEG - Binge Drink Days at 1 Month: LSEG - Binge Drink Days at 1 month
Arm/Group | GMI - Binge Drink Days at 1 Month | LSEG - Binge Drink Days at 1 Month
Number analyzed (Participants) | 89 | 82
Days | 3.0 [0.0 to 1.0] | 3.0 [0.0 to 3.0]

15. Primary Outcome: Binge Drink Days at 3 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days prior to 3-month follow-up. This measure represents the number of days the participant binge drank (5 or more standard drinks on a single day for males; 4 or more standard drinks on a single day for females) within the stated time period.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | GMI - Standard Ethanol Content Units (SECs) at 3 Months | LSEG - Standard Ethanol Content Units (SECs) at 3 Months
Number analyzed (Participants) | 87 | 77
Days | 5.1 [0.0 to 8.5] | 4.0 [0.0 to 3.5]

16. Primary Outcome: Binge Drink Days at 6 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 90 days prior to 6-month follow-up. This measure represents the number of days the participant binge drank (5 or more standard drinks on a single day for males; 4 or more standard drinks on a single day for females) within the stated time period.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Binge Drink Days at 6 Months: GMI - Binge Drink Days at 6 Months
- LSEG - Binge Drink Days at 6 Months: LSEG - Binge Drink Days at 6 Months
Arm/Group | GMI - Binge Drink Days at 6 Months | LSEG - Binge Drink Days at 6 Months
Number analyzed (Participants) | 85 | 75
Days | 6.2 [0.0 to 9.0] | 5.7 [0.0 to 9.7]

17. Primary Outcome: Illicit Drug Use Days at Baseline
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of drug use in the 30 days prior to Baseline. This measure represents the number of illicit drug use days within the stated time period.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Illicit Drug Use Days at Baseline: GMI - Illicit Drug Use Days at Baseline
- LSEG - Illicit Drug Use Days at Baseline: LSEG - Illicit Drug Use Days at Baseline
Arm/Group | GMI - Illicit Drug Use Days at Baseline | LSEG - Illicit Drug Use Days at Baseline
Number analyzed (Participants) | 93 | 91
Days | 6.2 [0.0 to 9.0] | 7.7 [0.0 to 14.0]

18. Primary Outcome: Illicit Drug Use Days at 1 Month
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 30 days prior to 1-month follow-up. This measure represents the number of illicit drug use days within the stated time period.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Illicit Drug Use Days at 1 Month: GMI - Illicit Drug Use Days at 1 month
- LSEG - Illicit Drug Use Days at 1 Month: LSEG - Illicit Drug Use Days at 1 month
Arm/Group | GMI - Illicit Drug Use Days at 1 Month | LSEG - Illicit Drug Use Days at 1 Month
Number analyzed (Participants) | 89 | 82
Days | 2.2 [0.0 to 1.0] | 1.7 [0.0 to 1.0]

19. Primary Outcome: Illicit Drug Use Days at 3 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 60 days prior to 3-month follow-up. This measure represents the number of illicit drug use days within the stated time period.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Illicit Drug Use Days at 3 Months: GMI - Illicit Drug Use Days at 3 months
- LSEG - Illicit Drug Use Days at 3 Months: LSEG - Illicit Drug Use Days at 3 months
Arm/Group | GMI - Illicit Drug Use Days at 3 Months | LSEG - Illicit Drug Use Days at 3 Months
Number analyzed (Participants) | 87 | 77
Days | 2.0 [0.0 to 1.0] | 2.5 [0.0 to 0.5]

20. Primary Outcome: Illicit Drug Use Days at 6 Months
Description: The Timeline Follow-Back (TLFB) calendar was used to assess retrospective self-report of alcohol in the 90 days prior to 6-month follow-up. This measure represents the number of illicit drug use days within the stated time period.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Days
Groups:
- GMI - Illicit Drug Use Days at 6 Months: GMI - Illicit Drug Use Days at 6 months
- LSEG - Illicit Drug Use Days at 6 Months: LSEG - Illicit Drug Use Days at 6 months
Arm/Group | GMI - Illicit Drug Use Days at 6 Months | LSEG - Illicit Drug Use Days at 6 Months
Number analyzed (Participants) | 85 | 75
Days | 3.4 [0.0 to 2.0] | 3.3 [0.0 to 1.7]

21. Primary Outcome: Substance Use Disorder Treatment Sessions at Baseline
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days prior to Baseline. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Substance Use Disorder Treatment Sessions at Baseline: GMI - Substance Use Disorder Treatment Sessions at Baseline
- LSEG - Substance Use Disorder Treatment Sessions at Baseline: LSEG - Substance Use Disorder Treatment Sessions at Baseline
Arm/Group | GMI - Substance Use Disorder Treatment Sessions at Baseline | LSEG - Substance Use Disorder Treatment Sessions at Baseline
Number analyzed (Participants) | 93 | 91
Sessions | 3.7 [0.0 to 5.0] | 4.7 [0.0 to 6.0]

22. Primary Outcome: Substance Use Disorder Treatment Sessions at 1 Month
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days prior to 1-month follow-up. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Substance Use Disorder Treatment Sessions at 1 Month: GMI - Substance Use Disorder Treatment Sessions at 1 month
- LSEG - Substance Use Disorder Treatment Sessions at 1 Month: LSEG - Substance Use Disorder Treatment Sessions at 1 month
Arm/Group | GMI - Substance Use Disorder Treatment Sessions at 1 Month | LSEG - Substance Use Disorder Treatment Sessions at 1 Month
Number analyzed (Participants) | 89 | 82
Sessions | 20.9 [0.0 to 40.0] | 22.2 [0.0 to 40.0]

23. Primary Outcome: Substance Use Disorder Treatment Sessions at 3 Months
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 60 days prior to 3-month follow-up. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Substance Use Disorder Treatment Sessions at 3 Months: GMI - Substance Use Disorder Treatment Sessions at 3 months
- LSEG - Substance Use Disorder Treatment Sessions at 3 Months: LSEG - Substance Use Disorder Treatment Sessions at 3 months
Arm/Group | GMI - Substance Use Disorder Treatment Sessions at 3 Months | LSEG - Substance Use Disorder Treatment Sessions at 3 Months
Number analyzed (Participants) | 87 | 77
Sessions | 8.1 [0.0 to 12.5] | 6.3 [0.0 to 8.5]

24. Primary Outcome: Substance Use Disorder Treatment Sessions at 6 Months
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 60 days prior to 6-month follow-up. Treatment sessions included the outpatient substance use disorder treatment group sessions and individual sessions.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Substance Use Disorder Treatment Sessions at 6 Months: GMI - Substance Use Disorder Treatment Sessions at 6 months
- LSEG - Substance Use Disorder Treatment Sessions at 6 Months: LSEG - Substance Use Disorder Treatment Sessions at 6 months
Arm/Group | GMI - Substance Use Disorder Treatment Sessions at 6 Months | LSEG - Substance Use Disorder Treatment Sessions at 6 Months
Number analyzed (Participants) | 85 | 75
Sessions | 3.2 [0.0 to 3.0] | 1.8 [0.0 to 2.0]

25. Primary Outcome: Twelve-Step Sessions Attended at Baseline
Description: A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 30 days prior to Baseline.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Twelve-Step Sessions Attended at Baseline: GMI - Twelve-Step Sessions Attended at Baseline
- LSEG - Twelve-Step Sessions Attended at Baseline: LSEG - Twelve-Step Sessions Attended at Baseline
Arm/Group | GMI - Twelve-Step Sessions Attended at Baseline | LSEG - Twelve-Step Sessions Attended at Baseline
Number analyzed (Participants) | 93 | 91
Sessions | 5.2 [0.0 to 6.0] | 3.8 [0.0 to 6.0]

26. Primary Outcome: Twelve-Step Sessions Attended at 1 Month
Description: A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 30 days prior to 1-month follow-up.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Twelve-Step Sessions Attended at 1 Month: GMI - Twelve-Step Sessions Attended at 1 month
- LSEG - Twelve-Step Sessions Attended at 1 Month: LSEG - Twelve-Step Sessions Attended at 1 month
Arm/Group | GMI - Twelve-Step Sessions Attended at 1 Month | LSEG - Twelve-Step Sessions Attended at 1 Month
Number analyzed (Participants) | 89 | 82
Sessions | 10.7 [0.0 to 19.0] | 10.8 [0.0 to 18.0]

27. Primary Outcome: Twelve-Step Sessions Attended at 3 Months
Description: A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended 60 days prior to 3-month follow-up.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Twelve-Step Sessions Attended at 3 Months: GMI - Twelve-Step Sessions Attended at 3 months
- LSEG - Twelve-Step Sessions Attended at 3 Months: LSEG - Twelve-Step Sessions Attended at 3 months
Arm/Group | GMI - Twelve-Step Sessions Attended at 3 Months | LSEG - Twelve-Step Sessions Attended at 3 Months
Number analyzed (Participants) | 87 | 77
Sessions | 9.8 [0.0 to 17.0] | 7.5 [0.0 to 13.5]

28. Primary Outcome: Twelve-Step Sessions Attended at 6 Months
Description: A Treatment Attendance Calendar was used to record the number of self-reported 12-step sessions attended in the 90 days prior to 6-month follow-up.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: Sessions
Groups:
- GMI - Twelve-Step Sessions Attended at 6 Months: GMI - Twelve-Step Sessions Attended at 6 months
- LSEG - Twelve-Step Sessions Attended at 6 Months: LSEG - Twelve-Step Sessions Attended at 6 months
Arm/Group | GMI - Twelve-Step Sessions Attended at 6 Months | LSEG - Twelve-Step Sessions Attended at 6 Months
Number analyzed (Participants) | 85 | 75
Sessions | 6.7 [0.0 to 9.7] | 3.8 [0.0 to 6.7]

29. Primary Outcome: Times Involved in Community Participation Activities at Baseline
Description: A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 30 days prior to Baseline.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: # of times activity completed
Groups:
- GMI - Times Involved in Community Participation Activities at: GMI - Times Involved in Community Participation Activities at Baseline
- LSEG - Times Involved in Community Participation Activities at: LSEG - Times Involved in Community Participation Activities at Baseline
Arm/Group | GMI - Times Involved in Community Participation Activities at | LSEG - Times Involved in Community Participation Activities at
Number analyzed (Participants) | 93 | 91
# of times activity completed | 10.4 [1.0 to 15.0] | 14 [2.0 to 19.0]

30. Primary Outcome: Times Involved in Community Participation Activities at 1 Month
Description: A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 30 days prior to 1-month follow-up.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: # of time activity completed
Groups:
- GMI - Times Involved in Community Participation Activities at: GMI - Times Involved in Community Participation Activities at 1 month
- LSEG - Times Involved in Community Participation Activities at: LSEG - Times Involved in Community Participation Activities at 1 month
Arm/Group | GMI - Times Involved in Community Participation Activities at | LSEG - Times Involved in Community Participation Activities at
Number analyzed (Participants) | 89 | 82
# of time activity completed | 18.4 [6.0 to 30.0] | 25.2 [7.0 to 40.0]

31. Primary Outcome: Times Involved in Community Participation Activities at 3 Months
Description: A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 60 days prior to 3-month follow-up.
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: # of times activity completed
Groups:
- GMI - Times Involved in Community Participation Activities at: GMI - Times Involved in Community Participation Activities at 3 months
- LSEG - Times Involved in Community Participation Activities at: LSEG - Times Involved in Community Participation Activities at 3 months
Arm/Group | GMI - Times Involved in Community Participation Activities at | LSEG - Times Involved in Community Participation Activities at
Number analyzed (Participants) | 87 | 77
# of times activity completed | 16.7 [3.5 to 23.5] | 19.4 [3.0 to 29.5]

32. Primary Outcome: Times Involved in Community Participation Activities at 6 Months
Description: A calendar was used to record the number of times a participant participated in an activity in the community (e.g. museum, library, baseball game) in the 90 days prior to 6-month follow-up.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: # of times activity completed
Groups:
- GMI - Times Involved in Community Participation Activities at: GMI - Times Involved in Community Participation Activities at 6 months
- LSEG - Times Involved in Community Participation Activities at: LSEG - Times Involved in Community Participation Activities at 6 months
Arm/Group | GMI - Times Involved in Community Participation Activities at | LSEG - Times Involved in Community Participation Activities at
Number analyzed (Participants) | 85 | 75
# of times activity completed | 16.7 [2.0 to 25.7] | 14.5 [2.0 to 26.0]

33. Primary Outcome: Days Involved in Productive Work Activities at Baseline
Description: A calendar was used to record the number of times a participant participated in a productive work activity (e.g. volunteered or worked at a job) in the 30 days prior to Baseline.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: # of days
Groups:
- GMI - Days Involved in Productive Work Activities at Baseline: GMI - Days Involved in Productive Work Activities at Baseline
- LSEG - Days Involved in Productive Work Activities at Baseline: LSEG - Days Involved in Productive Work Activities at Baseline
Arm/Group | GMI - Days Involved in Productive Work Activities at Baseline | LSEG - Days Involved in Productive Work Activities at Baseline
Number analyzed (Participants) | 93 | 91
# of days | 2.2 [0.0 to 1.0] | 3.0 [0.0 to 2.0]

34. Primary Outcome: Days Involved in Productive Work Activities at 1 Month
Description: A calendar was used to record the number of times a participant participated in a productive work activity (e.g. volunteered or worked at a job) in the 30 days prior to 1-month follow-up.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: # of days
Groups:
- GMI - Days Involved in Productive Work Activities at 1 Month: GMI - Days Involved in Productive Work Activities at 1 month
- LSEG - Days Involved in Productive Work Activities at 1 Month: LSEG - Days Involved in Productive Work Activities at 1 month
Arm/Group | GMI - Days Involved in Productive Work Activities at 1 Month | LSEG - Days Involved in Productive Work Activities at 1 Month
Number analyzed (Participants) | 89 | 82
# of days | 3.6 [0.0 to 3.0] | 3.5 [0.0 to 3.0]

35. Primary Outcome: Days Involved in Productive Work Activities at 3 Months
Description: A calendar was used to record the number of times a participant participated in a productive work activity (e.g. volunteered or worked at a job) in the 60 days prior to 3-month follow-up
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: # of days
Groups:
- GMI - Days Involved in Productive Work Activities at 3 Months: GMI - Days Involved in Productive Work Activities at 3 months
- LSEG - Days Involved in Productive Work Activities at 3 Months: LSEG - Days Involved in Productive Work Activities at 3 months
Arm/Group | GMI - Days Involved in Productive Work Activities at 3 Months | LSEG - Days Involved in Productive Work Activities at 3 Months
Number analyzed (Participants) | 87 | 77
# of days | 7.0 [0.0 to 13.5] | 7.0 [0.0 to 14.0]

36. Primary Outcome: Days Involved in Productive Work Activities at 6 Months
Description: A calendar was used to record the number of times a participant participated in a productive work activity (e.g. volunteered or worked at a job) in the 90 days prior to 6-month follow-up.
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: # of days
Groups:
- GMI - Days Involved in Productive Work Activities at 6 Months: GMI - Days Involved in Productive Work Activities at 6 months
- LSEG - Days Involved in Productive Work Activities at 6 Months: LSEG - Days Involved in Productive Work Activities at 6 months
Arm/Group | GMI - Days Involved in Productive Work Activities at 6 Months | LSEG - Days Involved in Productive Work Activities at 6 Months
Number analyzed (Participants) | 85 | 75
# of days | 8.0 [0.0 to 16.7] | 9.8 [0.0 to 22.0]

37. Secondary Outcome: Mental Health Treatment Sessions at Baseline
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days prior to Baseline. Treatment sessions included individual sessions with outpatient mental health staff.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Mental Health Treatment Sessions at Baseline: For those receiving GMI - Mental Health Treatment Sessions
- LSEG - Mental Health Treatment Sessions at Baseline: For those receiving LSEG - Mental Health Treatment Sessions
Arm/Group | GMI - Mental Health Treatment Sessions at Baseline | LSEG - Mental Health Treatment Sessions at Baseline
Number analyzed (Participants) | 93 | 91
sessions | 0.36 [0 to 0] | 0.20 [0 to 0]

38. Secondary Outcome: Mental Health Treatment Sessions at 1 Month
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 30 days prior to 1-month follow-up. Treatment sessions included individual sessions with outpatient mental health staff.
Time Frame: 1 Month
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Mental Health Treatment Sessions at 1 Month: For those receiving GMI - Mental Health Treatment Sessions at 1 Month
- LSEG - Mental Health Treatment Sessions at 1 Month: For those receiving LSEG - Mental Health Treatment Sessions at 1 Month
Arm/Group | GMI - Mental Health Treatment Sessions at 1 Month | LSEG - Mental Health Treatment Sessions at 1 Month
Number analyzed (Participants) | 89 | 82
sessions | 0.79 [0 to 1] | 0.39 [0 to 0]

39. Secondary Outcome: Mental Health Treatment Sessions at 3 Months
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 60 days prior to 3-month follow-up. Treatment sessions included individual sessions with outpatient mental health staff.
Time Frame: 3 Months
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Mental Health Treatment Sessions at 3 Months: For those receiving GMI - Mental Health Treatment Sessions at 3 Months
- LSEG - Mental Health Treatment Sessions at 3 Months: For those receiving LSEG - Mental Health Treatment Sessions at 3 Months
Arm/Group | GMI - Mental Health Treatment Sessions at 3 Months | LSEG - Mental Health Treatment Sessions at 3 Months
Number analyzed (Participants) | 87 | 77
sessions | 1.0 [0 to 1] | 0.25 [0 to 0]

40. Secondary Outcome: Mental Health Treatment Sessions at 6 Months
Description: A Treatment Attendance Calendar was used to record the number of objective treatment sessions documented in each participants VA Computerized Patient Record System for the 90 days prior to 6-month follow-up. Treatment sessions included individual sessions with outpatient mental health staff.
Time Frame: 6 Months
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Mental Health Treatment Sessions at 6 Months: For those receiving GMI - Mental Health Treatment Sessions at 6 Months
- LSEG - Mental Health Treatment Sessions at 6 Months: For those receiving LSEG - Mental Health Treatment Sessions at 6 Months
Arm/Group | GMI - Mental Health Treatment Sessions at 6 Months | LSEG - Mental Health Treatment Sessions at 6 Months
Number analyzed (Participants) | 85 | 75
sessions | 0.78 [0 to 0.70] | 0.27 [0 to 0]

41. Secondary Outcome: Substance Use Disorder and Mental Health Treatment Sessions at Baseline
Description: This specific measure combined the number substance use disorder treatment sessions and mental health treatment sessions attended for the 30 days prior to Baseline.
Time Frame: 30 days prior to Baseline
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI -Substance Use Disorder and Mental Health Treatment Sessio: For those receiving GMI - Substance Use Disorder and Mental Health Treatment Sessions at Baseline
- LSEG - Substance Use Disorder and Mental Health Treatment Sess: For those receiving LSEG - Substance Use Disorder and Mental Health Treatment Sessions at Baseline
Arm/Group | GMI -Substance Use Disorder and Mental Health Treatment Sessio | LSEG - Substance Use Disorder and Mental Health Treatment Sess
Number analyzed (Participants) | 93 | 91
sessions | 4.0 [0 to 5] | 4.9 [0 to 6]

42. Secondary Outcome: Substance Use Disorder and Mental Health Treatment Sessions at 1 Month
Description: This specific measure combined the number substance use disorder treatment sessions and mental health treatment sessions attended for the 30 days prior to 1-month follow-up.
Time Frame: 1 Month
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Substance Use Disorder and Mental Health Treatment Sessi: For those receiving GMI - Substance Use Disorder and Mental Health Treatment Sessions at 1 Month
- LSEG - Substance Use Disorder and Mental Health Treatment Sess: For those receiving LSEG - Substance Use Disorder and Mental Health Treatment Sessions at 1 Month
Arm/Group | GMI - Substance Use Disorder and Mental Health Treatment Sessi | LSEG - Substance Use Disorder and Mental Health Treatment Sess
Number analyzed (Participants) | 89 | 82
sessions | 21.7 [1 to 42] | 22.6 [1 to 41]

43. Secondary Outcome: Substance Use Disorder and Mental Health Treatment Sessions at 3 Months
Description: This specific measure combined the number substance use disorder treatment sessions and mental health treatment sessions attended for the 60 days prior to 3-month follow-up.
Time Frame: 3 Months
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Substance Use Disorder and Mental Health Treatment Sessi: For those receiving GMI - Substance Use Disorder and Mental Health Treatment Sessions at 3 Months
- LSEG - Substance Use Disorder and Mental Health Treatment Sess: For those receiving LSEG - Substance Use Disorder and Mental Health Treatment Sessions at 3 Months
Arm/Group | GMI - Substance Use Disorder and Mental Health Treatment Sessi | LSEG - Substance Use Disorder and Mental Health Treatment Sess
Number analyzed (Participants) | 87 | 77
sessions | 9.1 [0.5 to 13] | 6.5 [0 to 9]

44. Secondary Outcome: Substance Use Disorder and Mental Health Treatment Sessions at 6 Months
Description: This specific measure combined the number substance use disorder treatment sessions and mental health treatment sessions attended for the 90 days prior to 6-month follow-up.
Time Frame: 6 Months
Measure: Mean (Inter-Quartile Range); unit: sessions
Groups:
- GMI - Substance Use Disorder and Mental Health Treatment Sessi: For those receiving GMI - Substance Use Disorder and Mental Health Treatment Sessions at 6 Months
- LSEG - Substance Use Disorder and Mental Health Treatment Sess: For those receiving LSEG - Substance Use Disorder and Mental Health Treatment Sessions at 6 Months
Arm/Group | GMI - Substance Use Disorder and Mental Health Treatment Sessi | LSEG - Substance Use Disorder and Mental Health Treatment Sess
Number analyzed (Participants) | 85 | 75
sessions | 4.0 [0 to 3.67] | 2.0 [0 to 2.67]

45. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at Baseline for Alcohol Use
Description: The ASI-Lite will be used to measure addiction severity Min value:0 Max value: 1 Higher score indicates greater problem severity
Time Frame: 30 days prior to Baseline
Population: The ASI-Lite measures addiction severity
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for: GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for Alcohol Use
- LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline fo: LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline for Alcohol Use
Arm/Group | GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for | LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline fo
Number analyzed (Participants) | 90 | 88
score on a scale | 0.50 (.22) | 0.50 (.22)

46. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 1 Month for Alcohol Use
Description: as for outcome 45
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - ASI -- 1 Month Composite Score for Alcohol Use: GMI - ASI -- 1 month Composite Score for Alcohol Use
- LSEG - ASI -- 1 Month Composite Score for Alcohol Use: LSEG - ASI -- 1 month Composite Score for Alcohol Use
Arm/Group | GMI - ASI -- 1 Month Composite Score for Alcohol Use | LSEG - ASI -- 1 Month Composite Score for Alcohol Use
Number analyzed (Participants) | 84 | 67
score on a scale | 0.18 (0.23) | 0.19 (0.25)

47. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 3 Months for Alcohol Use
Description: as for outcome 45
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - ASI -- 3 Months Composite Score for Alcohol Use: GMI - ASI -- 3 months Composite Score for Alcohol Use
- LSEG - ASI -- 3 Months Composite Score for Alcohol Use: LSEG - ASI -- 3 months Composite Score for Alcohol Use
Arm/Group | GMI - ASI -- 3 Months Composite Score for Alcohol Use | LSEG - ASI -- 3 Months Composite Score for Alcohol Use
Number analyzed (Participants) | 81 | 66
score on a scale | 0.31 (0.35) | 0.27 (0.40)

48. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 6 Months for Alcohol Use
Description: as for outcome 45
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - ASI -- 6 Months Composite Score for Alcohol Use: GMI - ASI -- 6 months Composite Score for Alcohol Use
- LSEG - ASI -- 6 Months Composite Score for Alcohol Use: LSEG - ASI -- 6 months Composite Score for Alcohol Use
Arm/Group | GMI - ASI -- 6 Months Composite Score for Alcohol Use | LSEG - ASI -- 6 Months Composite Score for Alcohol Use
Number analyzed (Participants) | 76 | 72
score on a scale | 0.49 (0.57) | 0.41 (0.56)

49. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at Baseline for Psychiatric Status
Description: as for outcome 45
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for: GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for Psychiatric Status
- LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline fo: LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline for Psychiatric Status
Arm/Group | GMI - Addiction Severity Index-Lite (ASI-Lite) at Baseline for | LSEG - Addiction Severity Index-Lite (ASI-Lite) at Baseline fo
Number analyzed (Participants) | 89 | 86
score on a scale | 0.47 (0.21) | 0.40 (0.23)

50. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 1 Month for Psychiatric Status
Description: as for outcome 45
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Addiction Severity Index-Lite (ASI-Lite) at 1 Month for: GMI - Addiction Severity Index-Lite (ASI-Lite) at 1 month for Psychiatric Status
- LSEG - Addiction Severity Index-Lite (ASI-Lite) at 1 Month for: LSEG - Addiction Severity Index-Lite (ASI-Lite) at 1 month for Psychiatric Status
Arm/Group | GMI - Addiction Severity Index-Lite (ASI-Lite) at 1 Month for | LSEG - Addiction Severity Index-Lite (ASI-Lite) at 1 Month for
Number analyzed (Participants) | 71 | 71
score on a scale | 0.28 (0.26) | 0.26 (0.24)

51. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 3 Month for Psychiatric Status
Description: as for outcome 45
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Addiction Severity Index-Lite (ASI-Lite) at 3 Months for: GMI - Addiction Severity Index-Lite (ASI-Lite) at 3 months for Psychiatric Status
- LSEG - Addiction Severity Index-Lite (ASI-Lite) at 3 Month for: LSEG - Addiction Severity Index-Lite (ASI-Lite) at 3 months for Psychiatric Status
Arm/Group | GMI - Addiction Severity Index-Lite (ASI-Lite) at 3 Months for | LSEG - Addiction Severity Index-Lite (ASI-Lite) at 3 Month for
Number analyzed (Participants) | 79 | 60
score on a scale | 0.30 (0.28) | 0.26 (0.25)

52. Secondary Outcome: Addiction Severity Index-Lite (ASI-Lite) at 6 Months for Psychiatric Status
Description: as for outcome 45
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Addiction Severity Index-Lite (ASI-Lite) at 6 Months for: GMI - Addiction Severity Index-Lite (ASI-Lite) at 6 months for Psychiatric Status
- LSEG - Addiction Severity Index-Lite (ASI-Lite) at 6 Months fo: LSEG - Addiction Severity Index-Lite (ASI-Lite) at 6 months for Psychiatric Status
Arm/Group | GMI - Addiction Severity Index-Lite (ASI-Lite) at 6 Months for | LSEG - Addiction Severity Index-Lite (ASI-Lite) at 6 Months fo
Number analyzed (Participants) | 70 | 59
score on a scale | 0.38 (0.28) | 0.30 (0.26)

53. Secondary Outcome: Short Inventory of Problems (SIP) at Baseline
Description: Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Time Frame: 30 days prior to Baseline
Population: Short Inventory of Problems - Total Score at Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Short Inventory of Problems at Baseline - Total Score: GMI - Short Inventory of Problems Revised (SIP-R) at Baseline
- LSEG - Short Inventory of Problems Revised (SIP-R) at Baseline: LSEG - Short Inventory of Problems Revised (SIP-R) at Baseline
Arm/Group | GMI - Short Inventory of Problems at Baseline - Total Score | LSEG - Short Inventory of Problems Revised (SIP-R) at Baseline
Number analyzed (Participants) | 93 | 91
score on a scale | 27.0 (12.6) | 26.1 (12.2)

54. Secondary Outcome: Short Inventory of Problems at 1 Month
Description: Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Short Inventory of Problems Revised (SIP-R) at 1 Month: GMI - Short Inventory of Problems Revised (SIP-R) at 1 month
- LSEG - Short Inventory of Problems Revised (SIP-R) at 1 Month: LSEG - Short Inventory of Problems Revised (SIP-R) at 1 month
Arm/Group | GMI - Short Inventory of Problems Revised (SIP-R) at 1 Month | LSEG - Short Inventory of Problems Revised (SIP-R) at 1 Month
Number analyzed (Participants) | 89 | 82
score on a scale | 6.5 (10.6) | 6.9 (10.9)

55. Secondary Outcome: Short Inventory of Problems at 3 Months
Description: Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Short Inventory of Problems Revised (SIP-R) at 3 Months: GMI - Short Inventory of Problems Revised (SIP-R) at 3 months
- LSEG - Short Inventory of Problems Revised (SIP-R) at 3 Months: LSEG - Short Inventory of Problems Revised (SIP-R) at 3 months
Arm/Group | GMI - Short Inventory of Problems Revised (SIP-R) at 3 Months | LSEG - Short Inventory of Problems Revised (SIP-R) at 3 Months
Number analyzed (Participants) | 87 | 77
score on a scale | 9.8 (12.2) | 7.6 (10.7)

56. Secondary Outcome: Short Inventory of Problems at 6 Months
Description: Min value:0 Max value: 45 Higher score indicates higher number of consequences from alcohol and drug use
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Short Inventory of Problems Revised (SIP-R) at 6 Months: GMI - Short Inventory of Problems Revised (SIP-R) at 6 months
- LSEG - Short Inventory of Problems Revised (SIP-R) at 6 Months: LSEG - Short Inventory of Problems Revised (SIP-R) at 6 months
Arm/Group | GMI - Short Inventory of Problems Revised (SIP-R) at 6 Months | LSEG - Short Inventory of Problems Revised (SIP-R) at 6 Months
Number analyzed (Participants) | 85 | 75
score on a scale | 11.1 (12.4) | 10.8 (12.5)

57. Secondary Outcome: Social Support Survey Total Score at Baseline
Description: Min value:19 Max value:95 Higher score indicates higher support
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Social Support Survey Total Score at Baseline: GMI - Social Support Survey Total Score at Baseline
- LSEG - Social Support Survey Total Score at Baseline: LSEG - Social Support Survey Total Score at Baseline
Arm/Group | GMI - Social Support Survey Total Score at Baseline | LSEG - Social Support Survey Total Score at Baseline
Number analyzed (Participants) | 93 | 91
score on a scale | 61.1 (18.6) | 60.3 (21.2)

58. Secondary Outcome: Social Support Survey Total Score at 1 Month
Description: Min value:19 Max value:95 Higher score indicates higher support
Time Frame: 30 days prior to 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Social Support Survey Total Score at 1-month Follow-up: GMI - Social Support Survey Total Score at 1-month follow-up
- LSEG - Social Support Survey Total Score at 1-month Follow-up: LSEG - Social Support Survey Total Score at 1-month follow-up
Arm/Group | GMI - Social Support Survey Total Score at 1-month Follow-up | LSEG - Social Support Survey Total Score at 1-month Follow-up
Number analyzed (Participants) | 89 | 81
score on a scale | 63.3 (21) | 68.2 (20)

59. Secondary Outcome: Social Support Survey Total Score at 3 Months
Description: Min value:19 Max value:95 Higher score indicates higher support
Time Frame: 60 days prior to 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Social Support Survey Total Score at 3 Months: GMI - Social Support Survey Total Score at 3 months
- LSEG - Social Support Survey Total Score at 3 Months: LSEG - Social Support Survey Total Score at 3 months
Arm/Group | GMI - Social Support Survey Total Score at 3 Months | LSEG - Social Support Survey Total Score at 3 Months
Number analyzed (Participants) | 87 | 76
score on a scale | 63.1 (21.4) | 66.8 (19)

60. Secondary Outcome: Social Support Survey Total Score at 6 Months
Description: Min value:19 Max value:95 Higher score indicates higher support
Time Frame: 90 days prior to 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Social Support Survey Total Score at 6 Months: GMI - Social Support Survey Total Score at 6 months
- LSEG - Social Support Survey Total Score at 6 Months: LSEG - Social Support Survey Total Score at 6 months
Arm/Group | GMI - Social Support Survey Total Score at 6 Months | LSEG - Social Support Survey Total Score at 6 Months
Number analyzed (Participants) | 85 | 74
score on a scale | 61.2 (22) | 65.7 (19.2)

61. Secondary Outcome: Quality of Life Survey (QOLS) at Baseline
Description: Min value:16 Max value:112 Higher score indicates higher quality of life
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Quality of Life Survey (QOLS) at Baseline: GMI - Quality of Life Survey (QOLS) at Baseline
- LSEG - Quality of Life Survey (QOLS) at Baseline: LSEG - Quality of Life Survey (QOLS) at Baseline
Arm/Group | GMI - Quality of Life Survey (QOLS) at Baseline | LSEG - Quality of Life Survey (QOLS) at Baseline
Number analyzed (Participants) | 93 | 91
score on a scale | 61.6 (18.4) | 68.8 (17.6)

62. Secondary Outcome: Quality of Life Survey (QOLS) at 1 Month
Description: Min value:16 Max value:112 Higher score indicates higher quality of life
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Quality of Life Survey (QOLS) at 1 Month: GMI - Quality of Life Survey (QOLS) at 1 month
- LSEG - Quality of Life Survey (QOLS) at 1 Month: LSEG - Quality of Life Survey (QOLS) at 1 month
Arm/Group | GMI - Quality of Life Survey (QOLS) at 1 Month | LSEG - Quality of Life Survey (QOLS) at 1 Month
Number analyzed (Participants) | 89 | 81
score on a scale | 71.2 (15.3) | 73.5 (15.8)

63. Secondary Outcome: Quality of Life Survey (QOLS) at 3 Months
Description: Min value:16 Max value:112 Higher score indicates higher quality of life
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Quality of Life Survey (QOLS) at 3 Months: GMI - Quality of Life Survey (QOLS) at 3 months
- LSEG - Quality of Life Survey (QOLS) at 3 Months: LSEG - Quality of Life Survey (QOLS) at 3 months
Arm/Group | GMI - Quality of Life Survey (QOLS) at 3 Months | LSEG - Quality of Life Survey (QOLS) at 3 Months
Number analyzed (Participants) | 87 | 76
score on a scale | 72.4 (16.5) | 75.1 (17.9)

64. Secondary Outcome: Quality of Life Survey (QOLS) at 6 Months
Description: Min value:16 Max value:112 Higher score indicates higher quality of life
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Quality of Life Survey (QOLS) at 6 Months: GMI - Quality of Life Survey (QOLS) at 6 months
- LSEG - Quality of Life Survey (QOLS) at 6 Months: LSEG - Quality of Life Survey (QOLS) at 6 months
Arm/Group | GMI - Quality of Life Survey (QOLS) at 6 Months | LSEG - Quality of Life Survey (QOLS) at 6 Months
Number analyzed (Participants) | 85 | 75
score on a scale | 71.3 (18.3) | 72.6 (18.6)

65. Secondary Outcome: Brief Symptom Inventory (BSI-18) at Baseline
Description: Min value:0 Max value:72 Higher score indicates higher psychological distress
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Brief Symptom Inventory (BSI) at Baseline: GMI - Brief Symptom Inventory (BSI) at Baseline
- LSEG - Brief Symptom Inventory (BSI) at Baseline: LSEG - Brief Symptom Inventory (BSI) at Baseline
Arm/Group | GMI - Brief Symptom Inventory (BSI) at Baseline | LSEG - Brief Symptom Inventory (BSI) at Baseline
Number analyzed (Participants) | 93 | 91
score on a scale | 21.4 (14.0) | 19.3 (14.6)

66. Secondary Outcome: Brief Symptom Inventory(BSI-18) at 1 Month
Description: Min value:0 Max value:72 Higher score indicates higher psychological distress
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Brief Symptom Inventory (BSI) at 1 Month: GMI - Brief Symptom Inventory (BSI) at 1 month
- LSEG - Brief Symptom Inventory (BSI) at 1 Month: LSEG - Brief Symptom Inventory (BSI) at 1 month
Arm/Group | GMI - Brief Symptom Inventory (BSI) at 1 Month | LSEG - Brief Symptom Inventory (BSI) at 1 Month
Number analyzed (Participants) | 89 | 81
score on a scale | 15.9 (12.4) | 14.2 (12.6)

67. Secondary Outcome: Brief Symptom Inventory (BSI-18) at 3 Months
Description: Min value:0 Max value:72 Higher score indicates higher psychological distress
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Brief Symptom Inventory (BSI) at 3 Months: GMI - Brief Symptom Inventory (BSI) at 3 months
- LSEG - Brief Symptom Inventory (BSI) at 3 Months: LSEG - Brief Symptom Inventory (BSI) at 3 months
Arm/Group | GMI - Brief Symptom Inventory (BSI) at 3 Months | LSEG - Brief Symptom Inventory (BSI) at 3 Months
Number analyzed (Participants) | 87 | 76
score on a scale | 16.1 (13.8) | 13.1 (11.5)

68. Secondary Outcome: Brief Symptom Inventory (BSI-18) at 6 Months
Description: Min value:0 Max value:72 Higher score indicates higher psychological distress
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Brief Symptom Inventory (BSI) at 6 Months: GMI - Brief Symptom Inventory (BSI) at 6 months
- LSEG - Brief Symptom Inventory (BSI) at 6 Months: LSEG - Brief Symptom Inventory (BSI) at 6 months
Arm/Group | GMI - Brief Symptom Inventory (BSI) at 6 Months | LSEG - Brief Symptom Inventory (BSI) at 6 Months
Number analyzed (Participants) | 83 | 75
score on a scale | 17.2 (14.6) | 15.9 (13.6)

69. Secondary Outcome: SF-12 Health Survey Physical Summary Score at Baseline
Description: Physical summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Health Survey Physical Summary Score at Baseline: GMI - Health Survey Physical Summary Score at Baseline
- LSEG - Health Survey Physical Summary Score at Baseline: LSEG - Health Survey Physical Summary Score at Baseline
Arm/Group | GMI - Health Survey Physical Summary Score at Baseline | LSEG - Health Survey Physical Summary Score at Baseline
Number analyzed (Participants) | 89 | 88
score on a scale | 41.6 (11.8) | 41.6 (11.3)

70. Secondary Outcome: SF-12 Health Survey Physical Summary Score at 1 Month
Description: Physical summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Physical Summary Score at 1 Month: GMI - SF-12 Health Survey Physical Summary Score at 1 month
- LSEG - SF-12 Health Survey Physical Summary Score at 1 Month: LSEG - SF-12 Health Survey Physical Summary Score at 1 month
Arm/Group | GMI - SF-12 Health Survey Physical Summary Score at 1 Month | LSEG - SF-12 Health Survey Physical Summary Score at 1 Month
Number analyzed (Participants) | 86 | 78
score on a scale | 40.2 (11.4) | 43.6 (11.7)

71. Secondary Outcome: SF-12 Health Survey Physical Summary Score at 3 Months
Description: Physical summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Physical Summary Score at 3 Months: GMI - SF-12 Health Survey Physical Summary Score at 3 months
- LSEG - SF-12 Health Survey Physical Summary Score at 3 Months: LSEG - SF-12 Health Survey Physical Summary Score at 3 months
Arm/Group | GMI - SF-12 Health Survey Physical Summary Score at 3 Months | LSEG - SF-12 Health Survey Physical Summary Score at 3 Months
Number analyzed (Participants) | 85 | 71
score on a scale | 41.0 (10.5) | 42.2 (11.4)

72. Secondary Outcome: SF-12 Health Survey Physical Summary Score at 6 Months
Description: Physical summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Physical Summary Score at 6 Months: GMI - SF-12 Health Survey Physical Summary Score at 6 months
- LSEG - SF-12 Health Survey Physical Summary Score at 6 Months: LSEG - SF-12 Health Survey Physical Summary Score at 6 months
Arm/Group | GMI - SF-12 Health Survey Physical Summary Score at 6 Months | LSEG - SF-12 Health Survey Physical Summary Score at 6 Months
Number analyzed (Participants) | 80 | 74
score on a scale | 40.4 (11.1) | 40.8 (11.9)

73. Secondary Outcome: SF-12 Health Survey Mental Summary Score at Baseline
Description: Mental summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Mental Summary Score at Baseline: GMI - SF-12 Health Survey Mental Summary Score at Baseline
- LSEG - SF-12 Health Survey Mental Summary Score at Baseline: LSEG - SF-12 Health Survey Mental Summary Score at Baseline
Arm/Group | GMI - SF-12 Health Survey Mental Summary Score at Baseline | LSEG - SF-12 Health Survey Mental Summary Score at Baseline
Number analyzed (Participants) | 89 | 88
score on a scale | 35.9 (11.4) | 39.0 (11.9)

74. Secondary Outcome: SF-12 Health Survey Mental Summary Score at 1 Month
Description: Mental summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Mental Summary Score at 1 Month: GMI - SF-12 Health Survey Mental Summary Score at 1 month
- LSEG - SF-12 Health Survey Mental Summary Score at 1 Month: LSEG - SF-12 Health Survey Mental Summary Score at 1 month
Arm/Group | GMI - SF-12 Health Survey Mental Summary Score at 1 Month | LSEG - SF-12 Health Survey Mental Summary Score at 1 Month
Number analyzed (Participants) | 86 | 78
score on a scale | 43.9 (11.3) | 44.5 (10.8)

75. Secondary Outcome: SF-12 Health Survey Mental Summary Score at 3 Months
Description: Mental summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Mental Summary Score at 3 Months: GMI - SF-12 Health Survey Mental Summary Score at 3 months
- LSEG - SF-12 Health Survey Mental Summary Score at 3 Months: LSEG - SF-12 Health Survey Mental Summary Score at 3 months
Arm/Group | GMI - SF-12 Health Survey Mental Summary Score at 3 Months | LSEG - SF-12 Health Survey Mental Summary Score at 3 Months
Number analyzed (Participants) | 85 | 71
score on a scale | 43.0 (11.5) | 44.7 (10.5)

76. Secondary Outcome: SF-12 Health Survey Mental Summary Score at 6 Months
Description: Mental summary items are summed and weighed Min value:0 Max value:100 Higher score indicates higher level of health
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - SF-12 Health Survey Mental Summary Score at 6 Months: GMI - SF-12 Health Survey Mental Summary Score at 6 months
- LSEG - SF-12 Health Survey Mental Summary Score at 6 Months: LSEG - SF-12 Health Survey Mental Summary Score at 6 months
Arm/Group | GMI - SF-12 Health Survey Mental Summary Score at 6 Months | LSEG - SF-12 Health Survey Mental Summary Score at 6 Months
Number analyzed (Participants) | 80 | 74
score on a scale | 42.7 (11.8) | 44.6 (11.1)

77. Secondary Outcome: Treatment Motivation Questionnaire (TMQ) at Baseline
Description: The TMQ will be used to measure self-reported interest in attending treatment Scores within each subscale are averaged
  External:
  Min value:1 Max value:7 External:Higher score indicates higher external reasons for attending treatment (e.g.referred to treatment by legal system)
  Internal:
  Min value:1 Max value:7 Internal: Higher score indicates higher internal reasons for attending treatment (e.g. personal choice to attend treatment)
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Treatment Motivation Questionnaire (TMQ) at Baseline; LSEG - Treatment Motivation Questionnaire (TMQ) at Baseline: For those receiving GMI - The TMQ was used to assess self-reported interest in treatment at Baseline based on external reasons, internal reasons, help seeking and confidence.
Arm/Group | GMI - Treatment Motivation Questionnaire (TMQ) at Baseline | LSEG - Treatment Motivation Questionnaire (TMQ) at Baseline
Number analyzed (Participants) | 75 | 70
score on a scale
  External Reasons | 2.4 (1.2) | 2.6 (1.4)
  Internal Reasons | 6.1 (1.0) | 6.0 (0.9)

78. Secondary Outcome: Treatment Motivation Questionnaire (TMQ) at 1-month
Description: as for outcome 77
Time Frame: 30 days prior to 1-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Treatment Motivation Questionnaire (TMQ) at 1-month: Treatment Motivation Questionnaire (TMQ) at 1-month
- LSEG - Treatment Motivation Questionnaire (TMQ) at 1-month: LSEG - Treatment Motivation Questionnaire (TMQ) at 1-month
Arm/Group | GMI - Treatment Motivation Questionnaire (TMQ) at 1-month | LSEG - Treatment Motivation Questionnaire (TMQ) at 1-month
Number analyzed (Participants) | 76 | 68
score on a scale
  External Reasons | 2.2 (1.2) | 2.6 (1.5)
  Internal Reasons | 5.8 (1.1) | 5.8 (1.2)

79. Secondary Outcome: Treatment Motivation Questionnaire (TMQ) at 3-month
Description: as for outcome 77
Time Frame: 60 days prior to 3-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Treatment Motivation Questionnaire (TMQ) at 3-month: GMI - Treatment Motivation Questionnaire (TMQ) at 3-month
- LSEG - Treatment Motivation Questionnaire (TMQ) at 3-month: LSEG - Treatment Motivation Questionnaire (TMQ) at 3-month
Arm/Group | GMI - Treatment Motivation Questionnaire (TMQ) at 3-month | LSEG - Treatment Motivation Questionnaire (TMQ) at 3-month
Number analyzed (Participants) | 74 | 60
score on a scale
  External Reasons | 2 (1.2) | 2.5 (1.5)
  Internal Reasons | 5.4 (1.3) | 5.6 (1.3)

80. Secondary Outcome: Treatment Motivation Questionnaire (TMQ) at 6-months
Description: as for outcome 77
Time Frame: 90 days prior to 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Treatment Motivation Questionnaire (TMQ) at 6-month: GMI - Treatment Motivation Questionnaire (TMQ) at 6-month
- LSEG - Treatment Motivation Questionnaire (TMQ) at 6-month: LSEG - Treatment Motivation Questionnaire (TMQ) at 6-month
Arm/Group | GMI - Treatment Motivation Questionnaire (TMQ) at 6-month | LSEG - Treatment Motivation Questionnaire (TMQ) at 6-month
Number analyzed (Participants) | 68 | 52
score on a scale
  External Reasons | 2.2 (1.2) | 2.5 (1.2)
  Internal Reasons | 5.5 (1.2) | 5.3 (1.2)

81. Secondary Outcome: Fagerstrom Test for Nicotine Dependence at Baseline
Description: Min:0 Max:10 Higher score indicates higher level of nicotine dependence
Time Frame: 30 days prior to Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Fagerstrom Test for Nicotine Dependence at Baseline: GMI - Fagerstrom Test for Nicotine Dependence at Baseline
- LSEG - Fagerstrom Test for Nicotine Dependence at Baseline: LSEG - Fagerstrom Test for Nicotine Dependence at Baseline
Arm/Group | GMI - Fagerstrom Test for Nicotine Dependence at Baseline | LSEG - Fagerstrom Test for Nicotine Dependence at Baseline
Number analyzed (Participants) | 74 | 78
score on a scale | 4.5 (2.4) | 4.0 (2.2)

82. Secondary Outcome: Psychiatric Outpatient Satisfaction Scale - Total Score
Description: Min:13 Max:65 Higher score indicates better satisfaction
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - GMI - Psychiatric Outpatient Satisfaction Scale - Total: GMI - Psychiatric Outpatient Satisfaction Scale - Total Score
- LSEG - GMI - Psychiatric Outpatient Satisfaction Scale - Total: LSEG - GMI - Psychiatric Outpatient Satisfaction Scale - Total Score
Arm/Group | GMI - GMI - Psychiatric Outpatient Satisfaction Scale - Total | LSEG - GMI - Psychiatric Outpatient Satisfaction Scale - Total
Number analyzed (Participants) | 88 | 80
score on a scale | 61.1 (9.4) | 60.1 (9.8)

83. Secondary Outcome: Helping Alliance Questionnaire - Total Score
Description: Participant completed assessment on the final day of group and rated therapist based on their interactions over the 4 days.
  Min:19 Max:114 Higher score indicates stronger alliance with therapist
Time Frame: Completed during session 4 of treatment group (i.e. the final treatment session)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GMI - Helping Alliance Questionnaire - Total Score: GMI - Helping Alliance Questionnaire - Total Score
- LSEG - Helping Alliance Questionnaire - Total Score: LSEG - Psychiatric Outpatient Satisfaction Scale - Total Score
Arm/Group | GMI - Helping Alliance Questionnaire - Total Score | LSEG - Helping Alliance Questionnaire - Total Score
Number analyzed (Participants) | 78 | 77
score on a scale | 100.1 (10.9) | 101.6 (9.4)

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was collected through study completion, an average of 6 months.
Arm/Group | Group Motivational Interviewing (GMI) | Control Treatment Condition (CT)
All-Cause Mortality (participants affected / at risk) | 3/93 | 5/91
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/91
Other Adverse Events (participants affected / at risk) | 0/93 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02233738/Prot_SAP_000.pdf